CLINICAL TRIAL: NCT04490226
Title: Impact of Endogenous vs. Exogenous Ketone Bodies on Appetite Control and Macronutrient Oxidation
Brief Title: Endogenous vs. Exogenous Ketone Bodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anja Bosy-Westphal, Prof. Anja Bosy-Westphal, PhD, MD, University of Kiel
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ABW-2020-VK
Record Dates: First submitted 2020-07-16; First posted 2020-07-29 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: ketone bodies; appetite control; macronutrient oxidation; metabolic chamber; exogenous ketones
MeSH Terms: interventions — 3-Hydroxybutyric Acid; Exercise; Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: all subjects are undergoing each intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- fasting, active (Experimental): 36 hours fasting, PAL 1.6
  Interventions: Dietary Supplement: Beta-Hydroxybutyrate as Ca-Mg-salt, active; Dietary Supplement: ketogenic diet (KetoCal® 4:1 Neutral, Nutricia GmbH, Erlangen, Germany), active; Dietary Supplement: fasting, active; Dietary Supplement: fasting, inactive
- ketogenic diet, active (Experimental): 24 hours of ketogenic diet (liquid meals), PAL 1.6
  Interventions: Dietary Supplement: Beta-Hydroxybutyrate as Ca-Mg-salt, active; Dietary Supplement: ketogenic diet (KetoCal® 4:1 Neutral, Nutricia GmbH, Erlangen, Germany), active; Dietary Supplement: fasting, active; Dietary Supplement: fasting, inactive
- exogeneous ketone bodies, active (Experimental): 24 hours of ketone body supplements (Beta-Hydroxybutyrate as Ca-Mg-salt) additional to a normal diet (liquid meals), PAL 1.6
  Interventions: Dietary Supplement: Beta-Hydroxybutyrate as Ca-Mg-salt, active; Dietary Supplement: ketogenic diet (KetoCal® 4:1 Neutral, Nutricia GmbH, Erlangen, Germany), active; Dietary Supplement: fasting, active; Dietary Supplement: fasting, inactive
- fasting, inactive (Experimental): 36 hours fasting, PAL 1.3
  Interventions: Dietary Supplement: Beta-Hydroxybutyrate as Ca-Mg-salt, active; Dietary Supplement: ketogenic diet (KetoCal® 4:1 Neutral, Nutricia GmbH, Erlangen, Germany), active; Dietary Supplement: fasting, active; Dietary Supplement: fasting, inactive

INTERVENTIONS:
Dietary Supplement: Beta-Hydroxybutyrate as Ca-Mg-salt, active — 24 hour intervention with ketone body supplements additional to a normal diet (isocaloric diet in total) to induce ketosis (exogenous ketone bodies), in a metabolic chamber at physical activity level of 1.6, after one day of isocaloric diet in a metabolic chamber at physical activity level of 1.6.
Dietary Supplement: ketogenic diet (KetoCal® 4:1 Neutral, Nutricia GmbH, Erlangen, Germany), active — 24 hour interventions with ketogenic isocaloric diet to induce ketosis (endogenous ketone bodies), in a metabolic chamber at physical activity level of 1.6, after one day of isocaloric diet in a metabolic chamber at physical activity level of 1.6.
Dietary Supplement: fasting, active — 36 hours of fasting, in a metabolic chamber at physical activity level of 1.6, after one day of isocaloric diet in a metabolic chamber at physical activity level of 1.6.
Dietary Supplement: fasting, inactive — 36 hours of fasting, in a metabolic chamber at physical activity level of 1.3, after one day of isocaloric diet in a metabolic chamber at physical activity level of 1.3.
  The same intervention is reproduced one week later.

SUMMARY:
Aim of the study is to compare the origin of ketone bodies: endogenous ketone bodies due to 36 hours fasting or 24 hours of ketogenic diet vs. exogenous ketone bodies as supplements additional to normal diet.

Secondary aim of the study is to validate the new metabolic chambers.

DETAILED DESCRIPTION:
Each study week starts with a 3-day run-in period with controlled diet at home and ends with a test-meal (breakfast) in the lab and following food record over the rest of the day at home.

1. week: physical activity level (PAL) 1.3, 3 intervention days in the metabolic chamber: ad libitum energy intake, washout day, isocaloric diet, 36 hours fasting
2. week: physical activity level (PAL) 1.3, 2 intervention days in the metabolic chamber: isocaloric diet, 36 hours fasting
3. week: physical activity level (PAL) 1.6, 2 intervention days in the metabolic chamber: ad libitum energy intake, 36 hours fasting
4. week: physical activity level (PAL) 1.6, 2 intervention days in the metabolic chamber: isocaloric diet, ketogenic diet (isocaloric)
5. week: physical activity level (PAL) 1.6, 2 intervention days in the metabolic chamber: isocaloric diet, isocaloric diet + ketone body supplements (isocaloric)

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI 19-29 kg/m2
* low-medium habitual physical activity
* women using hormonal contraceptive

Exclusion Criteria:

* smoking
* chronic illnesses
* food allergies / intolerances
* vegans and vegetarians
* regular high physical activity (exercise >1 hour/d)
* current weight loss diet / weight loss of >5 kg in the last 3 months
* pregnant / lactating women
* persons incapable of giving informed legal consent

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
appetite control - ghrelin | 24 hours
  ghrelin concentration in plasma (24 hour AUC)
appetite control - GLP-1 concentration in plasma | 24 hours
  Glucose Like Peptide-1 concentration in plasma (24 hour AUC)
appetite control - PYY concentration in plasma | 24 hours
  Peptide YY concentration in plasma (24 hour AUC)
appetite control - subjective feelings of hunger | 24 hours
  measured with visual analogue scales (24 hour AUC). The scale consists of a 10 cm vertical line anchored with "not hungry at all" at the left side and with "extremely hungry" at the right side.
appetite control - satiety quotient | 30 min
  satiety quotient of standard test-breakfast after 24 hours of intervention

SECONDARY OUTCOMES:
macronutrient oxidation | 24 hours
  measured with indirect calorimetry in a metabolic chamber
energy expenditure | 24 hours
  measured with indirect calorimetry in a metabolic chamber
glycemia - glucose AUC | 24 hours
  glucose AUC from continuous glucose monitoring data
repeatability of energy expenditure measurements | 24 hours
  repeated measurement of 24h-energy expenditure in a metabolic chamber on inactive isocaloric and fasting days
ß-Hydroxybutyrate concentration in serum | 24 hours
  24 hour ß-Hydroxybutyrate concentration in serum (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, PhD, MD, Principal Investigator — Institute of Human Nutrition, Kiel University
Locations (1):
- Institute of Human Nutrition, Kiel, Germany

REFERENCES:
- [Derived] Hagele FA, Dorner R, Koop J, Lubken M, Seidel U, Rimbach G, Muller MJ, Bosy-Westphal A. Impact of one-day fasting, ketogenic diet or exogenous ketones on control of energy balance in healthy participants. Clin Nutr ESPEN. 2023 Jun;55:292-299. doi: 10.1016/j.clnesp.2023.03.025. Epub 2023 Apr 10. PMID 37202059
- [Derived] Dorner R, Hagele FA, Koop J, Rising R, Foerster T, Olsen T, Hasler M, Muller MJ, Bosy-Westphal A. Validation of energy expenditure and macronutrient oxidation measured by two new whole-room indirect calorimeters. Obesity (Silver Spring). 2022 Sep;30(9):1796-1805. doi: 10.1002/oby.23527. Epub 2022 Aug 4. PMID 35927795